CLINICAL TRIAL: NCT00497835
Title: Epilepsy Alert Device - Epilert Performance
Brief Title: Study of Algorithm for Epilepsy Alert Device
Status: Completed | Type: Observational
Sponsor: Biolert (Industry)
Responsible Party: Prof. Uri Kramer. Chief scientist, Biolert LTD
Other Study IDs: Biolert LTD
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2007-07

CONDITIONS: Motor Seizures
Keywords: motor seizures; accelerometer; algorithm; detection; alert
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: no Biospecimen
Oversight: Data Monitoring Committee: Yes

SUMMARY:
An accelerometer with transmitting ability is worn on the wrist. Data of movements during seizures will be analyzed to upgrade algorithm that will identify seizures.

DETAILED DESCRIPTION:
Patients undergoing Video-EEG telemetry will wear movement sensor on their wrist. The sensor will transmit continuous data to a laptop. Seizures' data (tonic or clonic) will be analyzed and transformed into an algorithm (up-graded existing preliminary algorithm).

In the second phase the algorithm will need to identify seizure events within one minute of the onset.

Both specificity ("false positive") and sensitivity ("false negative) will be than calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Long Term Monitoring for motor seizures

Exclusion Criteria:

* Invasive recording
* Psychogenic seizures

Ages: 1 Day to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to Video-LTM Unit with motor seizures.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2007-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Swetlana Kiperwasser, M.D., Principal Investigator — Tel-Aviv Sourasky Medical Center